CLINICAL TRIAL: NCT07282470
Title: Epigenetic Profiling and Liquid Biopsy: Perspectives for Personalized Medicine in Meningioma Patients
Brief Title: Epigenetic Profiling and Liquid Biopsy: Perspectives for Personalized Medicine in Meningioma Patients - MIND
Acronym: MIND
Status: Recruiting | Type: Observational
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Collaborators: University of Milan (Other); Università degli Studi del Piemonte Orientale Amedeo Avogadro (Other)
Responsible Party: Sponsor
Other Study IDs: MIND
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-12

CONDITIONS: Meningioma; Meningioma of Brain
Keywords: Meningioma; Machine Learning
MeSH Terms: conditions — Meningioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Tessuti FFPE, siero, plasma, EVs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective Cohort: 150 patients operated for non-recurrent meningioma between 2008 and 2016.
- Prospective Cohort: 60 patients diagnosed with meningioma recruited prospectively.

SUMMARY:
Meningiomas are the most common primary intracranial tumors. Current treatment relies on surgical resection and radiotherapy, but molecular predictors for recurrence are lacking. This study aims to investigate epigenetic features, specifically histone post-translational modifications (PTMs) and DNA methylation, to stratify patients. The study involves a retrospective cohort to define an epigenetic signature and a prospective cohort to validate it in tissues and liquid biopsies (plasma/EVs).

DETAILED DESCRIPTION:
The study is shaped by two phases. The first is a histone PTMs analysis in solid tissues from a retrospective cohort of 150 meningioma FFPE samples. The second step consists of validating the epigenetic signature in a prospective cohort of patients (n=60). The study addresses four main objectives: 1) Dissecting the informative power of epigenetic signatures (histone PTMs by MS) in tissues; 2) Validating signatures in prospective tissues and matched sera (circulating nucleosomes); 3) Assessing DNA methylation profiles from plasma-derived Extracellular Vesicles (EVs); 4) Developing a Machine Learning model integrating epi-proteomics, DNA-methylation, and clinical data for prognostic subtyping.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria (Retrospective & Prospective):

* Patient aged 18 years or older.
* First diagnosis of uni-focal meningioma of the convexity.
* Macroscopical total resection (Simpson 1-3).

(Retrospective only):

* Surgery performed between 2007 and 2016;
* availability of FFPE sample and medical records.

Exclusion Criteria:

* Genetic syndromes.
* Diffuse Meningeal Meningiomatosis.
* Patients who underwent experimental treatment in neo-adjuvant setting.

(Prospective only):

* Previous surgical/medical treatment for another meningioma;
* positive oncological history (e.g., breast cancer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Meningioma
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Definition of a novel epigenetic signature based on MS-profiling | Months 1-12
  Identification of histone post-translational modifications (PTMs) patterns in FFPE tissue samples capable of classifying tumor recurrence.

SECONDARY OUTCOMES:
Validation of epigenetic signature in prospective tissues | Months 13-18
  Validation of the histone PTMs signature using Mass Spectrometry on FFPE samples from the prospective cohort.
Validation of epigenetic biomarkers in circulating nucleosomes | Months 13-20
  Profiling histone PTMs in circulating nucleosomes from patient sera matching the tissues profiled.
DNA methylation profiling in plasma-EVs | Months 10-20
  Assessment of genome-wide DNA methylation profile from DNA extracted from plasma-derived Extracellular Vesicles.
Development of a Machine Learning prognostic classifier | Months 18-24
  Integration of epi-proteomics data, DNA-methylation profiles, and clinico-pathological information to predict recurrence.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Italy

IPD SHARING:
Plan to Share IPD: No